CLINICAL TRIAL: NCT00082563
Title: A Phase II, Randomized, Comparative Trial Of Azithromycin In Combination With Chloroquine Versus Chloroquine In The Eradication Of Asymptomatic Plasmodium Falciparum Infection In Semi-Immune Adults
Brief Title: Azithromycin in Combination With Chloroquine Versus Chloroquine in the Eradication of Asymptomatic Plasmodium Falciparum
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0661121
Record Dates: First submitted 2004-05-12; First posted 2004-05-14 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2011-04

CONDITIONS: Malaria, Falciparum
MeSH Terms: conditions — Malaria, Falciparum | interventions — Azithromycin; Chloroquine

INTERVENTIONS:
Drug: Azithromycin/Chloroquine
Drug: Chloroquine

SUMMARY:
The purpose of this study is to determine if Azithromycin in combination with chloroquine is superior to chloroquine alone in eradicating P. falciparum asexual parasitemia in asymptomatic, semi-immune adults in Western Kenya.

DETAILED DESCRIPTION:
The trial was terminated prematurely 9 November 2004 due to the inability to recruit the planned number of subjects. There were no safety or efficacy concerns regarding the study in the decision to terminate the trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult: male or female
* Asymptomatic mono-infection with P. falciparum parasitemia with a parasite density of 1000 - 30,000 parasites/Î¼L
* Age 18 years to 60 years
* Willingness to sign and ability to understand consent form
* Willingness and ability to return for scheduled follow up visits

Exclusion Criteria:

* Mixed malaria infection by Giemsa smear
* History of allergy to or hypersensitivity to chloroquine, Azithromycin or other macrolides (e.g. erythromycin, clarithromycin)
* Any of the following: a.) Antimalarial therapy administered in the past 4 weeks, including quinine therapy or an artemisinin derivative; or b.) An antibacterial with known antimalarial activity (including, erythromycin, doxycycline, clindamycin, cotrimoxazole) within one week prior to enrollment into the study
* Fever, history of fever in past 48 hours, or signs/symptoms of malaria (including acute or subacute headache, nausea, or vomiting)
* Inability to swallow oral medication
* Laboratory evidence or history of significant cardiovascular, liver, hematologic or renal functional abnormality
* Any situation which could prevent the patient from returning to follow up visits
* Pregnancy or breast feeding
* Any other concurrent illness that may confound the result
* Any other condition or circumstance that in the opinion of the Investigator may pose a threat to the study participant or study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2004-08; Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Parasite clearance

SECONDARY OUTCOMES:
tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer